CLINICAL TRIAL: NCT00983463
Title: Relative Abundance and Spatial Distribution of Lipids and Proteins in Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: Abundance and Distribution of Lipids and Proteins in Nonalcoholic Fatty Liver Disease (NAFLD)
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Charles R. Flynn, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: IRB #090657
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Nonalcoholic fatty liver disease (NAFLD); Nonalcoholic steatohepatitis (NASH); Obesity; Lipidomics; Proteomics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — liver biopsy, blood, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Obese, bariatric surgery, liver biopsy: Obese subjects approved and scheduled for bariatric surgery at Vanderbilt University Medical Center
- Normal BMI, abdominal surgery, liver biopsy: Normal weight subjects having elective abdominal surgery at Vanderbilt University Medical Center.
- Liver transplantation donors and recipients: All livers made available for implantation or explantation will be eligible.

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common type of liver disease in the United States. The incidence of NAFLD is very similar to that of obesity, type 2 diabetes, and the metabolic syndrome. The investigators hypothesize that there may be a relationship between over-nutrition, decreased physical activity and the development of fatty liver. The purpose of this study is to identify the types of fats and proteins, and the quantity of each, that are associated with increased severity of NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year of age
* Undergoing elective abdominal or bariatric surgery
* May have normal or elevated ALT/AST levels

Exclusion Criteria:

* Presence of viral hepatitis
* Significant alcohol use
* Intercurrent infections
* Use of any thiazolidinediones

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects having bariatric surgery or elective abdominal surgery at Vanderbilt University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2009-10; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
To identify and relatively quantify, using high performance liquid chromatography electrospray ionization mass spectrometry, select lipids and proteins present in human liver biopsies. | 2 years
To spatially profile, using matrix assisted laser desorption ionization time of flight mass spectrometry, select lipids and proteins present in human liver biopsies. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Flynn, PhD, Principal Investigator — Vanderbilt University Medical Center; Najji Abumrad, MD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Garcia AE, Kasim N, Tamboli RA, Gonzalez RS, Antoun J, Eckert EA, Marks-Shulman PA, Dunn J, Wattacheril J, Wallen T, Abumrad NN, Flynn CR. Lipoprotein Profiles in Class III Obese Caucasian and African American Women with Nonalcoholic Fatty Liver Disease. PLoS One. 2015 Nov 23;10(11):e0142676. doi: 10.1371/journal.pone.0142676. eCollection 2015. PMID 26599819